CLINICAL TRIAL: NCT01205022
Title: Phase I Trial of Radioimmunotherapy (Y-90 M5A) in Combination With FOLFIRI and Bevacizumab Chemotherapy for Metastatic Colorectal Carcinoma
Brief Title: Radiolabeled Monoclonal Antibody Therapy, Combination Chemotherapy, and Bevacizumab in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10038; NCI-2010-01962
Record Dates: First submitted 2010-09-16; First posted 2010-09-20 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Irinotecan; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes, leucovorin calcium IV over 2 hours, fluorouracil IV continuously over 46-48 hours, and bevacizumab IV over 30-90 minutes once every 2 weeks. Patients also receive yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A IV over 25 minutes once in weeks 3 and 9.Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: irinotecan hydrochloride; Drug: leucovorin calcium; Drug: fluorouracil; Biological: bevacizumab; Radiation: yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; camptothecin-11; CPT-11; irinotecan; U-101440E
Drug: leucovorin calcium — Given IV
  Other Names: calcium folinate; CF; CFR; citrovorum factor; LV; Wellcovorin
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU; Adrucil; Efudex; FU
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; anti-VEGF rhuMAb; Avastin; rhuMAb VEGF
Radiation: yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A — Given IV
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can find tumor cells and either kill them or carry tumor-killing substances to them without harming normal cells. Giving radioactive substances together with antibodies may be effective treatment for some advanced cancers. Drugs used in chemotherapy, such as irinotecan hydrochloride, fluorouracil, and leucovorin calcium (FOLFIRI), work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving radiolabeled monoclonal antibodies together with combination chemotherapy and bevacizumab may be an effective treatment for colorectal cancer.

PURPOSE: This phase I trial is studying the side effects, best way to give, and best dose of yttrium Y 90 DOTA anti-CEA (Carcinoembryonic antigen) monoclonal antibody M5A when given together with combination chemotherapy and bevacizumab in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the maximum tolerated dose of a combination of FOLFIRI chemotherapy, and intravenous yttrium-90 (90Y) M5A anti-CEA antibody.

SECONDARY OBJECTIVES:I. To study the progression free survival and response rate of this combined treatment in patients with stage IV colorectal cancer.II. To evaluate the biodistribution, clearance and metabolism of 90Y and 111In (indium-111) M5A administered intravenously.

OUTLINE: This is a dose-escalation study of yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A. Patients receive irinotecan hydrochloride IV over 90 minutes, leucovorin calcium IV over 2 hours, fluorouracil IV continuously over 46-48 hours, and bevacizumab IV over 30-90 minutes once every 2 weeks. Patients also receive yttrium Y 90 DOTA anti-CEA monoclonal antibody M5A IV over 25 minutes once in weeks 3 and 9. Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a Karnofsky performance status of > 60%
* Patients must have histological confirmation of colorectal carcinoma with stage IV disease or with unresectable disease
* Patients must have colorectal tumors that produce CEA as documented by either immunohistochemistry or by an elevated serum CEA
* Prior radiotherapy, immunotherapy, or chemotherapy must have been completed no less than 28 days prior to patient entry on this study and patients must have recovered from all acute expected side effects of the prior therapy. For patients who have undergone port placement, study treatment initiation must be at least 7 days post port placement
* Adequate bone marrow function as evidenced by hemoglobin > 10 g/dL, WBC > 4000/ul, an absolute granulocyte count of > 1,500/mm^3, and platelets > 150,000/ul; patients may be transfused to reach a hemoglobin > 10 g/dL
* In the dose-escalation phase, patients may have had a history of a prior malignancy; for the dose-expansion cohort, patients may have history of prior malignancy for which they have been disease free for five years with the exception of basal or squamous cell skin cancers or carcinoma in situ of the cervix
* Patients must have a total bilirubin < 1.5 mg/dL and a serum creatinine of < 2.0 mg/dL
* If a patient has previously received antibody, then serum anti-antibody testing must be negative
* Serum HIV testing and hepatitis B surface antigen and C antibody testing must be negative
* Women of childbearing potential must have a negative serum pregnancy test prior to entry and while on study must be practicing an effective form of contraception
* Patients must have measurable disease as defined by the modified RECIST criteria

Exclusion Criteria:

* Patients who have received radiation therapy to greater than 50% of their bone marrow
* Patients with any nonmalignant intercurrent illness (example cardiovascular, pulmonary, or central nervous system disease) that is either poorly controlled with currently available treatment or that is of such severity that the investigators deem it unwise to enter the patient on protocol shall be ineligible
* Patients with > 2+ protein by dipstick should undergo a 24 hour urine collection; patients with > 1gram proteinuria/ 24 hours are not eligible
* Patients may have received neoadjuvant and/or adjuvant chemotherapy and/or radiotherapy and present to the study in relapse; otherwise, no prior therapy is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of yttrium-90 (90Y) M5A anti-CEA antibody when given in combination with FOLFIRI chemotherapy and bevacizumab | 1 year post treatment

SECONDARY OUTCOMES:
Progression-free survival | 2 years post treatment
Overall survival | 2 years post treatment
Response rates | 2 years post treatment
Biodistribution, clearance, and metabolism of Y-90 and In-111-M5A | At baseline, 1 hour, and 4 hours post start of infusion and at scan times at 1 day, 2 days, 3-5 days, and 6-7 days post antibody infusion
Estimation of radiation doses to whole body, normal organs, and tumor through serial nuclear imaging | At 1-3 hours post start of antibody infusion, 1 day, 2 days, 3-5 days, and 6-7 days post antibody infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wong, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States